CLINICAL TRIAL: NCT04468347
Title: 18F-AV-1451 PET Imaging in the Preclinical, Prodromal and Dementia Phases of Alzheimer's Disease
Brief Title: Flortaucipir PET Imaging in the Preclinical, Prodromal and Dementia Phases of Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A08
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Alzheimer's disease (AD) (Experimental): Alzheimer's disease subjects receiving a flortaucipir PET scan at baseline and 12 months
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- Mild cognitive impairment (MCI) (Experimental): Mild cognitive impairment subjects receiving a flortaucipir PET scan at baseline and 12 months
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- Subjective memory complainers (SMC) (Experimental): Subjective memory complainers receiving a flortaucipir PET scan at baseline and 12 months
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- Cognitively normal (CN) (Experimental): Cognitively normal subjects receiving a flortaucipir PET scan at baseline and 12 months
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan

INTERVENTIONS:
Drug: Flortaucipir F18 — IV injection, 240 megabecquerel (MBq) (6.5 mCi)
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748; Tauvid
Procedure: Brain PET scan — positron emission tomography (PET) scan of the brain

SUMMARY:
A Phase 1 study designed to evaluate imaging characteristics of flortaucipir in the preclinical, prodromal and dementia phases of Alzheimer's disease.

DETAILED DESCRIPTION:
The Australian Imaging Biomarkers and Lifestyle Study (AIBL) is a multicenter multidisciplinary study of Alzheimer's disease and aging funded by the Commonwealth Scientific and Industrial Research Organisation (CSIRO) Flagship Initiative, involving research centers in both Victoria and Western Australia. The goal of the A08 protocol was to further investigate the positron emission tomography (PET) imaging results with flortaucipir in patients across the AD spectrum from individuals with subjective memory complaints (SMC) to those with dementia, based on recruitment into the parent AIBL study.

ELIGIBILITY:
Inclusion Criteria:

* Meet all inclusion criteria for the AIBL study protocol, with amyloid PET conducted or planned and MRI available
* Subjects in the MCI and AD groups required to have a reliable caregiver capable of providing information about the subjects' symptoms

Exclusion Criteria:

* lifetime history of schizophrenia, schizoaffective disorder, or bipolar disorder
* history of electroconvulsive therapy
* MRI contraindicated
* claustrophobic or, otherwise, unable to tolerate the imaging procedure
* current clinically significant cardiovascular disease or clinically significant abnormalities on screening electrocardiogram
* history of additional risk factors for Torsades de Pointes
* current clinically significant infectious disease, endocrine or metabolic disease, or pulmonary, renal, or hepatic impairment that the investigator believes would affect study participation
* history of cancer (other than skin or in situ prostate cancer) within the previous 5 years
* current drug or alcohol abuse/dependence
* history of alcohol abuse/dependence with 2 years of the onset of the symptoms of dementia
* females of childbearing potential who were not surgically sterile, not refraining from sexual activity, or not using reliable methods of contraception

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals, Inc.

REFERENCES:
- See also: Link to the Australian Imaging, Biomarker & Lifestyle Flagship Study of Ageing (AIBL) website — http://aibl.csiro.au/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between Oct 2014 and Feb 2018 from the Australian Imaging, Biomarker & Lifestyle Flagship Study of Ageing (AIBL)
Period: Overall Study
Arm/Group | Alzheimer's Disease (AD) | Mild Cognitive Impairment (MCI) | Subjective Memory Complainers (SMC) | Cognitively Normal (CN)
Started | 6 | 11 | 47 | 25
Baseline Flortacuipir PET Scan | 5 | 11 | 45 | 25
Completed | 4 | 10 | 41 | 21
Not Completed | 2 | 1 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alzheimer's Disease (AD) | Mild Cognitive Impairment (MCI) | Subjective Memory Complainers (SMC) | Cognitively Normal (CN) | Total
Number analyzed (Participants) | 5 | 11 | 45 | 25 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.2 (6.53) | 74.3 (5.82) | 77 (7.43) | 72.9 (4.67) | 75.4 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 26 | 13 | 45
  Male | 3 | 7 | 19 | 12 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 11 | 45 | 25 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 11 | 44 | 25 | 85
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 11 | 45 | 25 | 86
Mini Mental Status Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 22.6 (3.21) | 25.5 (2.84) | 28 (1.66) | 28.6 (0.99) | 27.5 (2.35)

OUTCOME MEASURES:

1. Primary Outcome: Flortaucipir PET Imaging (Quantitative)
Description: Flortaucipir PET cortical weighted average standardized uptake value ratio (SUVr). For SUVr, a value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline scan
Population: Inclusion in this analysis required that the subject's flortaucipir scan was analyzable for SUVr (1 AD, 1 MCI, 5 SMC, and 3 CN were not analyzable)
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVr)
Groups:
- Objectively Impaired: Combined AD and MCI group
- Non-objectively Compared: Combined SMC and CN groups
Arm/Group | Alzheimer's Disease (AD) | Mild Cognitive Impairment (MCI) | Objectively Impaired | Subjective Memory Complainers (SMC) | Cognitively Normal (CN) | Non-objectively Compared
Number analyzed (Participants) | 4 | 10 | 14 | 40 | 22 | 62
standardized uptake value ratio (SUVr) | 1.31 (0.059) | 1.13 (0.033) | 1.15 (0.031) | 1.08 (0.016) | 1.04 (0.028) | 1.07 (0.015)
Statistical Analysis 1: Comparison: Objectively Impaired vs Non-objectively Compared; Test type: Other; p < 0.0001, ANOVA; The two-way ANOVA included cognitive and amyloid status, and their interaction as fixed effects; Mean Difference (Net) = 0.16, Standard Error of Mean 0.038
Statistical Analysis 2: Comparison: Objectively Impaired vs Subjective Memory Complainers (SMC); Test type: Other; p = 0.0005, ANOVA; The two-way ANOVA included cognitive and amyloid status, and their interaction as fixed effects; Mean Difference (Net) = 0.14, Standard Error of Mean 0.038
Statistical Analysis 3: Comparison: Subjective Memory Complainers (SMC) vs Cognitively Normal (CN); Test type: Other; p = 0.2161, ANOVA; The two-way ANOVA included cognitive and amyloid status, and their interaction as fixed effects; Mean Difference (Net) = -0.04, Standard Error of Mean 0.033

2. Primary Outcome: Number of Participants With Advanced AD Pattern Flortaucipir PET Scan and Relationship to Cognitive Status
Description: Scans were visually read independently by two expert readers at the sponsor, blinded to any clinical information. Subject scans were categorized as follows: Advanced AD Scan Pattern (τAD++), Moderate AD Scan Pattern (τAD+), Not AD Scan Pattern (τAD-). For this analysis, subjects with Advanced (τAD++) scans were analyzed vs. the combined Moderate and Not AD pattern groups (τAD+/τAD-). Amyloid status was obtained by florbetapir or carbon-11-labeled Pittsburgh compound B ([C-11] PiB) PET results available from the parent AIBL study.
Time Frame: baseline scan
Population: Rows display flortaucipir scan results by subjects who were amyloid positive and amyloid negative at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Alzheimer's Disease (AD) | Mild Cognitive Impairment (MCI) | Subjective Memory Complainers (SMC) | Cognitively Normal (CN)
Number analyzed (Participants) | 5 | 11 | 45 | 25
Participants
  Amyloid Positive: number analyzed (Participants) | 4 | 5 | 20 | 4
  Amyloid Positive: Advanced AD Scan Pattern (τAD++) | 2 | 3 | 9 | 0
  Amyloid Positive: Not Advanced AD Pattern | 2 | 2 | 11 | 4
  Amyloid Negative: number analyzed (Participants) | 1 | 6 | 25 | 21
  Amyloid Negative: Advanced AD Scan Pattern (τAD++) | 1 | 0 | 3 | 1
  Amyloid Negative: Not Advanced AD Pattern | 0 | 6 | 22 | 20
Statistical Analysis 1: Comparison: Alzheimer's Disease (AD) vs Mild Cognitive Impairment (MCI) vs Subjective Memory Complainers (SMC) vs Cognitively Normal (CN); Test type: Other; p = 0.1998, Cochran-Mantel-Haenszel

3. Primary Outcome: Number of Participants With AD Pattern Flortaucipir PET Scan and Relationship to Cognitive Status
Description: Scans were visually read independently by two expert readers at the sponsor, blinded to any clinical information. Subject scans were categorized as follows: Advanced AD Scan Pattern (τAD++), Moderate AD Scan Pattern (τAD+), Not AD Scan Pattern (τAD-). For this analysis, subjects with AD Pattern scans (Advanced [τAD++] and Moderate [τAD+] Scan Pattern) were combined vs. the Not AD pattern group (τAD-). Amyloid status was obtained by florbetapir or carbon-11-labeled Pittsburgh compound B ([C-11] PiB) PET results available from the parent AIBL study.
Time Frame: baseline scan
Population: Rows display flortaucipir scan results by subjects who were amyloid positive and amyloid negative at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Alzheimer's Disease (AD) | Mild Cognitive Impairment (MCI) | Subjective Memory Complainers (SMC) | Cognitively Normal (CN)
Number analyzed (Participants) | 5 | 11 | 45 | 25
Participants
  Amyloid Positive: number analyzed (Participants) | 4 | 5 | 20 | 4
  Amyloid Positive: AD Pattern Scan (Advanced or Moderate) | 2 | 4 | 11 | 0
  Amyloid Positive: Not AD Pattern Scan | 2 | 1 | 9 | 4
  Amyloid Negative: number analyzed (Participants) | 1 | 6 | 25 | 21
  Amyloid Negative: AD Pattern Scan (Advanced or Moderate) | 1 | 0 | 6 | 1
  Amyloid Negative: Not AD Pattern Scan | 0 | 6 | 19 | 20
Statistical Analysis 1: Comparison: Alzheimer's Disease (AD) vs Mild Cognitive Impairment (MCI) vs Subjective Memory Complainers (SMC) vs Cognitively Normal (CN); Test type: Other; p = 0.0646, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: End of study for AE reporting was 48 hours after flortaucipir administration at each imaging visit.
Description: Adverse Events were defined as occurring or worsening after injection of dose, within 48 hours post injection, at an imaging visit. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to flortaucipir.
Arm/Group | Alzheimer's Disease (AD) | Mild Cognitive Impairment (MCI) | Subjective Memory Complainers (SMC) | Cognitively Normal (CN)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11 | 0/45 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/11 | 0/45 | 0/25
Other Adverse Events (participants affected / at risk) | 0/5 | 0/11 | 1/45 | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alzheimer's Disease (AD) (N=5) | Mild Cognitive Impairment (MCI) (N=11) | Subjective Memory Complainers (SMC) (N=45) | Cognitively Normal (CN) (N=25)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-02-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT04468347/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04468347/SAP_001.pdf